CLINICAL TRIAL: NCT05270941
Title: Platelet Rich Fibrin Prepared With Titanium Connective Tissue Graft in Treatment of Gingival Recessions
Brief Title: Platelet-Rich Fibrin Prepared With Titanium in the Treatment of Multiple Gingival Recessions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Dilek Özkan Şen, dr. öğr. üyesi, Necmettin Erbakan University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: dilek özkan şen
Record Dates: First submitted 2022-02-12; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Gingival Recession
Keywords: recession; gingival; subepithelial connective tissue graft
MeSH Terms: conditions — Gingival Recession | interventions — Titanium

STUDY DESIGN:
Intervention Model Description: As a randomized controlled clinical trial, in the patients' bilateral recession sites, while gingival recessions of one group were treated with T-PRF, the gingival recessions of the other group were treated with SCTG using a simple randomization method.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Groups (Active Comparator): Control groups. This clinical trial was designed as a split-mouth, randomized, controlled clinical trial. Bilateral gingival recession defects were randomly assigned to the test (CAF+T-PRF) or control (CAF+SCTG) groups after initially evaluating the clinical parameters and randomized by coin flip method.
  Intervention: Procedure: Control groups
  Interventions: Procedure: COMPARISON OF PLATELET-RICH FIBRIN PREPARED WITH TITANIUM AND SUBEPITHELIAL CONNECTIVE TISSUE GRAFT
- Test Group (Experimental): Test groups. This clinical trial was designed as a split-mouth, randomized, controlled clinical trial. Bilateral gingival recession defects were randomly assigned to the test (CAF+T-PRF) or control (CAF+SCTG) groups after initially evaluating the clinical parameters and randomized by coin flip method.
  Intervention: Procedure: Control groups Intervention: Procedure: test groups
  Interventions: Procedure: COMPARISON OF PLATELET-RICH FIBRIN PREPARED WITH TITANIUM AND SUBEPITHELIAL CONNECTIVE TISSUE GRAFT

INTERVENTIONS:
Procedure: COMPARISON OF PLATELET-RICH FIBRIN PREPARED WITH TITANIUM AND SUBEPITHELIAL CONNECTIVE TISSUE GRAFT — In the study, 118 maxillary bilateral multiple Miller Class I gingival recessions in 20 patients were treated. The gingival recessions were randomly treated with either T-PRF (58 teeth) or SCTG (60 teeth) using the modified coronally positioned flap technique. Gingival index, plaque index, probing pocket depth, gingival thickness, recession height, recession width, keratinized gingival width, and open root surface area were measured and recorded at baseline and at the 6th month. Postoperative pain levels were evaluated using the VAS (Visual Analogue Scale), and healing status was evaluated using the wound healing index. The pre- and post-treatment results of both treatment groups and the differences between the groups were evaluated and compared.
  Other Names: MODİFİYE CORONALLY ADVANCED FLAP

SUMMARY:
The aim of this study was to treat the areas with Miller Class I bilateral multiple gingival recession in the maxillary teeth using the Titanium Platelet-Rich Fibrin (T-PRF), an autogenous biomaterial applied in combination with a Modified Coronally Positioned Flap (MCPF) prepared using microsurgical techniques, and the gold standard Subepithelial Connective Tissue Graft (SCTG), to evaluate the efficacy of the treatments and to compare the clinical results 6 months after the treatment.

DETAILED DESCRIPTION:
AİM:

The aim of this study was to treat the areas with Miller Class I bilateral multiple gingival recession in the maxillary teeth using the Titanium Platelet-Rich Fibrin (T-PRF), an autogenous biomaterial applied in combination with a Modified Coronally Positioned Flap (MCPF) prepared using microsurgical techniques, and the gold standard Subepithelial Connective Tissue Graft (SCTG), to evaluate the efficacy of the treatments and to compare the clinical results 6 months after the treatment.

MATERIALS AND METHODS A total of 20 patients (118 defects), consisting of 13 females and 7 males, with maxillary bilateral Miller Class I gingival recession who were aged between 18 and 65, applied to Necmettin Erbakan University, Faculty of Dentistry, Department of Periodontology and had aesthetic anxiety and sensitivity problems due to multiple gingival recessions were included in our study. As a randomized controlled clinical trial, in the patients' bilateral recession sites, while gingival recessions of one group were treated with T-PRF, the gingival recessions of the other group were treated with SCTG using a simple randomization method. The study protocol was in accordance with the Declaration of Helsinki of 1975, as revised in 2002 and was submitted to and approved by the ethical committee of Necmettin Erbakan University and the Ministry of Health General Directorate of Health Services (protocol number:2019/238). All patients included in the study were given detailed information about the clinical trial, and their written informed consent was obtained. The study was performed between January 2019 and November 2020 in Necmettin Erbakan University Department of Periodontology.

The individuals were divided into 2 groups in accordance with the study protocol:

Group1: SCTG group (n=60) Group2: T-PRF group (n=58) The criteria for inclusion in the study were determined as systemically and periodontally healthy volunteers between the ages of 18-65, the absence of parafunctional habits, non-smoking, the presence of Miller Class I gingival recession defect in teeth located in the bilateral maxillary region, the absence of any hard tissue defects in the relevant region and the absence of a restorative, endodontic procedure or periodontal surgical intervention, a full-mouth plaque score (FMPS) of ≤ 25%, having a marginal gingival thickness of at least 1 mm in the area with gingival recession, the absence of a shallow hard palate dome, having a soft tissue thickness of at least 3 mm, the absence of torus in the area where the graft was taken, the absence of any systemic disease, not using antibiotics for any reason in the last 6 months, the presence of at least 20 teeth in the mouth, not being pregnant and breastfeeding, and patients who applied to the periodontology clinic with various periodontal problems and were indicated for connective tissue graft operation due to gingival recession. The individuals who were outside the exclusion criteria and did not agree to participate in the study were excluded from the study.

In the study with a sample size of 118, the effect size value (G * Power 3.1 for Windows) calculated based on the power (1-β err probe) = 95% and α = 5% t-test was determined as 0.334 for the analysis of repeated measurements.

ELIGIBILITY:
Inclusion Criteria:

* The criteria for inclusion in the study were determined as systemically and periodontally healthy volunteers between the ages of 18-65,
* the absence of parafunctional habits, non-smoking
* the presence of Miller Class I gingival recession defect in teeth located in the bilateral maxillary region
* the absence of any hard tissue defects in the relevant region and the absence of a restorative, endodontic procedure or periodontal surgical intervention
* a full-mouth plaque score (FMPS) of ≤ 25%
* having a marginal gingival thickness of at least 1 mm in the area with gingival recession
* the absence of a shallow hard palate dome
* having a soft tissue thickness of at least 3 mm
* the absence of torus in the area where the graft was taken
* the absence of any systemic disease
* not using antibiotics for any reason in the last 6 months
* the presence of at least 20 teeth in the mouth
* not being pregnant and breastfeeding, and patients who applied to the periodontology clinic with various periodontal problems and were indicated for connective tissue graft operation due to gingival recession

Exclusion Criteria:

* The individuals who were outside the exclusion criteria and did not agree to participate in the study were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-01-12 (Actual); Primary Completion 2020-11-29 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Complete root coverage [ Time Frame: 6 months | 6 MONTHS
  Change from baseline in gingival recession was be assessed at 1, and 6 months.
Gingival recession depth [ Time Frame: 6 months ] | 6 months.
  Change from baseline in gingival recession was be assessed at 6 months

SECONDARY OUTCOMES:
Keratinized tissue width [ Time Frame: 6 months ] | 6 months.
  Change from baseline in keratinized tissue at 6 months.
Pain scores [ Time Frame: first week after operations ] | first week
  Pain level evaluated on visual analog scale

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Necmettin Erbakan Üniversitesi Diş Hekimliği Fakültesi, Konya, Meram
  - Necmettin Erbakan Üniversitesi Diş Hekimliği Fakültesi, Konya

IPD SHARING:
Plan to Share IPD: Undecided